CLINICAL TRIAL: NCT06855121
Title: The Norwegian Immunotherapy in Multiple Myeloma Study - A Population-based Longitudinal Observational Multicenter Study on Effectiveness and Complications of Immunotherapy in Multiple Myeloma in the Norwegian Myeloma Cohort
Brief Title: The Norwegian Immunotherapy in Multiple Myeloma Study
Acronym: NIMMS
Status: Recruiting | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); Haukeland University Hospital (Other); Helse Stavanger HF (Other Government); Oslo University Hospital (Other); University Hospital, Akershus (Other); Sykehuset i Vestfold Hospital Trust (Unknown); University Hospital of North Norway (Other); Ålesund Hospital, Norway (Unknown); Helse Nord-Trøndelag HF (Other); Sorlandet Hospital HF (Other Government); Førde Hospital Trust (Other); Molde Hospital (Other); Bodø Hospital, Norway (Unknown); Helse Fonna (Other); Volda Hospital (Other); Diakonhjemmet Hospital (Other); Telemark Hospital Trust (Unknown); Kristiansund Hospital (Other); Vestre Viken Hospital Trust (Other); Lovisenberg Diakonale Hospital (Other); Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor
Other Study IDs: NIMMS
Record Dates: First submitted 2025-01-24; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Myeloma Multiple; Plasma Cell Leukemia; AL Amyloidosis
Keywords: bispesific antibodies; teclistamab; elranatamab; talquetamab; cilta-cel; ide-cel; ciltacabtagene autoleucel; idecabtagene vicleucel; CRS; ICAN; infections; supportive care
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Plasma Cell; Immunoglobulin Light-chain Amyloidosis; Infections | interventions — talquetamab; idecabtagene vicleucel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and bone marrow (in responding patients), nasopharyngeal secretion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Teclistamab — Real-world use and dosing
Drug: Elranatamab — Real-world use and dosing
Biological: Ciltacabtagene Autoleucel — Real-world use.
Drug: Talquetamab — Real-world use and dosing
Biological: Idecabtagene vicleucel — Real-world use and dosing

SUMMARY:
The goal of this observational study is to study the effectiveness and complications of novel immunotherapies used in the treatment of multiple myeloma in routine care in Norway. The aim is to close knowledge gaps, generate evidence for future clinical trials and contribute to future consensus on how to monitor for adverse events, and what mitigation strategies should be implemented, so that we can increase patient survival and quality-of-life.

ELIGIBILITY:
Inclusion criteria

* Participants age ≥ 18 years
* Prior diagnosis of one of the following

  * Multiple myeloma as defined according to IMWG criteria
  * Primary plasma cell leukemia as defined according to IMWG consensus definition
  * AL-amyloidosis as defined according to IMWG criteria
* Planned treatment with one of the following outside clinical trials (list to be amended based on approvals within the EU):

  * Teclistamab (Tecvayli)
  * Elranatamab (Elrexfio)
  * Talquetamab (Talvey)
  * Idecabtagene vicleucel (ide-cel/Abecma)
  * Ciltacabtagene autoleucel (cilta-cel/Carvykti)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multiple myeloma, plasma cell leukemia or AL amyloidosis treated at study sites outside clinical trials.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2037-12-01 (Estimated)

PRIMARY OUTCOMES:
Determine the real-world overall response rates (ORR) | From date of treatment start and until date of first documented progression or start of next line of therapy, whichever came first, assessed up to ten years.
Determine real-world progression-free survival (PFS) | From date of treatment start and until date of first documented progression or death, whichever came first, , assessed up to ten years.
Determine real-world time-to-next treatment (TTNT) | From date of treatment start and until date of start of next treatment, assessed up to ten years.
Determine real-world overall survival (OS) | From date of treatment start and until death, assessed up to ten years.
Describe the frequency and grading of adverse events of special interest (AESI), defined as described below. | From date of treatment start until the date of start of next line of treatment or death, whichever came first, assessed up to 10 years
  * Cytokine release syndrome (CRS) (ASTCT grade 1-5),
  * Infections (CTCAE grade 1-5)
  * Neurological adverse events (including, but not limited to, ICANS, peripheral sensory and/or motor neuropathy, neurocognitive and hypokinetic movement disorder) (CTCAE 5.0. grade 1-5).
  * Immune effector cell-associated hematotoxicity (ICAHT) (EHA/EBMT Consensus Grading 1-4)27
  * Secondary malignancies, dysgeusia, skin- and nail adverse events, pain, hemophagocytic lymphohistiocytosis (HLH) and tumor lysis syndrome (CTCAE grade 1-5)
Frequency and grading of all other adverse events occurring during treatment according to CTCAE 5.0 (only grade 3 or higher will be reported). | From start of treatment and until start of next treatment or death, assessed up to ten years.
Describe the microbiological pattern (positive cultures/PCR) of infections during treatment. | From start of treatment and start of next treatment line or death, assessed up to ten years.
Describe the antibiotic resistance pattern of positive cultures. | From start of treatment and start of next treatment line or death, assessed up to ten years.
Describe the prevalence of common airway viruses during treatment and at end-of-treatment. | From date of start of treatment and until end of treatment, assessed up to ten years.
Determine the real-world use of antimicrobial prophylaxis (antibiotics, antivirals, vaccines, immunoglobulines) before and during therapy. | From enrollment and until end of treatment, assessed up to ten years.

CONTACTS AND LOCATIONS:
Locations (23):
- Norway (23):
  - Sørlandet Hospital - Arendal, Arendal
  - Ålesund hospital, Department of hematology, Ålesund
  - Haukeland University Hospital, Bergen
  - Bodø Hospital, Bodø
  - Bærum Hospital, Bærum
  - Drammen hospital, Drammen
  - Førde hospital, Førde
  - Innlandet hospital trust, Gjøvik
  - Haugesund hospital, Haugesund
  - Sørlandet hospital, Kristiansand
  - Nordmøre and Romsdal Hospital - Kristiansund, Kristiansund
  - Levanger hospital, Levanger
  - Nordmøre and Romsdal Hospital - Molde, Molde
  - Akershus University Hospital (AHUS), Nordbyhagen
  - Diakonhjemmet hospital, Oslo
  - Lovisenberg Diaconal Hospital, Oslo
  - Oslo Myeloma Center, Oslo University Hospital, Oslo
  - Telemark Hospital Trust, Skien
  - Stavanger University hospital, Stavanger
  - University hospital of North Norway, Tromsø
  - St. Olavs hospital HF, Trondheim
  - Vestfold Hospital Trust, Tønsberg
  - Volda hospital, Volda

IPD SHARING:
Plan to Share IPD: No